CLINICAL TRIAL: NCT05447845
Title: A Novel Rapid, Reproducible and Accurate Computerized Visual Acuity Test
Brief Title: Rapid Computerized Visual Acuity Test
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Eytan Z Blumenthal, MD, Head of the Department of Ophthalmology, Rambam Health Care Campus
Other Study IDs: 0163-17-RMB
Record Dates: First submitted 2022-06-11; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Vision Disorders; Refractive Errors; Retinal Disease; Cataract; Corneal Disease
MeSH Terms: conditions — Vision Disorders; Refractive Errors; Retinal Diseases; Cataract; Corneal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy: healthy volunteers with no known ocular condition
  Interventions: Diagnostic Test: Computerized visual acuity assessment program
- Patients: Subjects with diseases of the eye or the orbit
  Interventions: Diagnostic Test: Computerized visual acuity assessment program

INTERVENTIONS:
Diagnostic Test: Computerized visual acuity assessment program — Each subject underwent visual acuity assessments using the Early Treatment Diabetic Retinopathy Study (ETDRS) chart and the computerized program

SUMMARY:
A novel computerized visual acuity test was developed and tested on both healthy persons and patients with ocular conditions. Visual acuity outcomes of the computerized test will be compared to the Early Treatment Diabetic Retinopathy Study (ETDRS) in measures of reproducibility, accuracy and numbers of questions.

ELIGIBILITY:
Inclusion Criteria:

- age 18 years old and older

Exclusion Criteria:

* visual acuity <0.2 decimal for the patient group
* visual acuity <0.5 decimal for the healthy group

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * healthy volunteers with no known ocular condition or past ocular surgery for the healthy group.
  * patients with ocular conditions who presented for treatment at the Department of Ophthalmology at the Outpatient Clinic at Rambam Health Care Campus
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | through study completion, an average of 1 year
  visual acuity was displayed in decimal units in the computerized program and by the number of letters in the early treatment diabetic retinopathy study chart (ETDRS).

CONTACTS AND LOCATIONS:
Overall Officials: Eytan Z Blumenthal, MD, Principal Investigator — Head of the Department of Ophthalmology
Locations (1):
- Department of Ophthalmology at Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No
The data collected is relevant to the computerized software developed by the team, the software is currently not available for other researchers' use. Therefore, sharing IPD will not be of further investigational importance to researchers out of the study team.

REFERENCES:
- [Background] Mimouni M, Shamir RR, Cohen AD, El-Yaniv R, Cohen MJ, Joskowicz L, Blumenthal EZ. A Comparison of different scoring terminations rules for visual acuity testing: from a computer simulation to a clinical study. Curr Eye Res. 2019 Jul;44(7):790-795. doi: 10.1080/02713683.2019.1589524. Epub 2019 Apr 8. PMID 30829080
- [Background] Cohen ADN, Mimouni M, El-Yaniv R, Blumenthal EZ. Shortening the Early Treatment Diabetic Retinopathy Study visual acuity test utilizing a novel computer software: reproducibility in control and patient eyes. Acta Ophthalmol. 2021 Dec;99(8):e1281-e1288. doi: 10.1111/aos.14807. Epub 2021 Mar 19. PMID 33742567